CLINICAL TRIAL: NCT05078554
Title: HPV Vaccination (Human Papilloma Virus), or How to Address Male Homosexuality in General Practice in Alsace?
Brief Title: HPV and Male Homosexuality in General Practice?
Acronym: HPV
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8048
Record Dates: First submitted 2021-10-13; First posted 2021-10-14 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2021-10

CONDITIONS: Papilloma Viral Infection
Keywords: Papilloma Viral Infection; HPV; HPV vaccine
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to find out whether young MSM (men who have sex with men) believe it is important for their GP to be informed of their sexual orientation, in order to improve their clinical, especially with HPV vaccination.

The secondary objective is to analyze the state of knowledge about the HPV vaccine and the value of HPV vaccine in this target population.

ELIGIBILITY:
Inclusion criteria:

* Age: 18-26 years
* Consultation at the HUS Cegidd as part of an STI screening
* Subject who expressed no opposition to participating in the study

Exclusion criteria:

* Refusal of the patient to participate in the study
* Subject who had already benefited from HPV vaccination (at least one dose)
* Inability to give informed consent
* Subject under safeguarde of justice
* Subject under guardianship or under curatorship

Ages: 18 Years to 26 Years | Sex: Male
Age Groups: Adult
Study Population: Subjetc aged between 18-26 years consulting at the HUS Cegidd as part of an STI screening
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
Retrospective descriptive study of vaccination against HPV (Human Papilloma Virus) in Alsace? | Files analysed retrospectively from April 27, 2021 to January 27, 2020 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service du Trait d'Union - Hôpitaux Universitaires de Strasbourg, Strasbourg, France